CLINICAL TRIAL: NCT01648309
Title: Neuropsychological Testing in Patients Undergoing TAVI
Brief Title: Neuropsychological Testing in Patients Undergoing Transvascular Aortic Valve Implantation
Acronym: TAVIPSYCH
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ronen Leker, Director - Stroke Center, Hadassah Medical Organization
Other Study IDs: TAVIPSYCH-HMO-CTIL; TAVI registry Hadassah; TAVI registry Hadassah (Registry Identifier: TAVI HADASSAH)
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; TAVI; neuropsychological; cognitive; candidates for TAVI
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAVI: patients with significant aortic stenosis that are candidates for transvascular aortic valve implantation
  Interventions: Other: Neuropsychological testing

INTERVENTIONS:
Other: Neuropsychological testing — This is an observational study

SUMMARY:
The purpose of this study is to examine the neuropsychological effects of transvascular aortic valve implantation (TAVI). Patients undergoing TAVI usually suffer from congestive heart failure and low cardiac output which may limit their cognitive abilities. TAVI results in significant improvements in cardiac function and therefore may improve cognitive functions. However, TAVI may also be associated with stroke and may therefore have a negative impact on cognition. Therefore, in this study the investigators wish to perform a battery of standardized neuropsychological tests before and after TAVI to test the net effects of TAVI on cognitive performance over time.

The investigators plan to include all patients planned to have TAVI in the study and to test them before, 3,7, 30 and 360 days post TAVI with a standardized battery of test.

ELIGIBILITY:
Inclusion Criteria:

* All patients with severe aortic stenosis that are candidates for TAVI
* Able to perform the testing
* Able to sign informed consent

Exclusion Criteria:

* Language barriers precluding the administration of the testing
* Existing dementia
* Existing disease limiting life expectancy to less than 180 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with severe aortic stenosis that are candidates for TAVI
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
net change in neuropsychological tests between baseline and day 180 from TAVI | 180 days
  The study will assess changes in cognitive performance between baseline (prior to TAVI) and 180 days after TAVI

SECONDARY OUTCOMES:
net difference between cognitive measures before TAVI and at day 30 after TAVI | 30 days
  The study will evaluate net differences between scores obtained on cognitive tests at baseline prior to TAVI and day 30 after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Ronen R Leker, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel